CLINICAL TRIAL: NCT01626014
Title: Making End of Life Decision in Ovarian Cancer: When to Enter Hospice? A Prototype Interactive Computer Program for Patients and Providers
Brief Title: Interactive Educational Website for Women With Ovarian Cancer & Caregivers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012NTLS005
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Stage III Ovarian Cancer; Stage IV Ovarian Cancer; Recurrent Ovarian Cancer; Fallopian Tube Cancer
Keywords: Stage III ovarian cancer; Stage IV ovarian cancer; recurrent ovarian cancer; primary peritoneal cancer; fallopian tube cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Using the Prototype System website: An interactive educational system for patients and their caregivers includes features allowing users to create their own profile, share a journal with others, and post to respective discussion forums. In addition, core intervention components include distress monitoring, educational items, details about the healthcare team and an areas to keep track of questions for providers.
  Interventions: Behavioral: Prototype System
- Control Group (Active Comparator): Using the Usual Care Educational Website : a website which will contain information regarding ovarian cancer however it will not be interactive. It will contain pdf documents of the material handed out in clinic (usual care).
  Interventions: Behavioral: Usual Care Educational Website

INTERVENTIONS:
Behavioral: Usual Care Educational Website — Using the control website: Participants access a website with standard ovarian cancer informational handouts.
  Arms: Control Group
Behavioral: Prototype System — An interactive system for patients and their caregivers includes features allowing users to create their own profile, share a journal with others, and post to respective discussion forums. In addition, core intervention components include distress monitoring, educational items, details about the healthcare team and an areas to keep track of questions for providers.
  Arms: Intervention Group

SUMMARY:
Ovarian cancer accounts for more deaths than any other gynecologic malignancy. The majority of patients are diagnosed with Stage III-IV disease. Nearly 80% of these patients will recur resulting in 5-year survival rates of 14-32%. Although enrollment is increasing in hospice, hospice programs have been challenged to reach eligible patients. Several factors limit the number of people who enroll in hospice and the length of their hospice stay. Prognostication challenges and the increasing availability of cancer therapies for people with cancer set the stage for a mismatch between certification of a 6 month prognosis and contemporary medical care. Additionally patients often are not aware of hospice and the services they can provide.

DETAILED DESCRIPTION:
In this study, we will pilot-test a technology-based approach for women with Stage III/IV or recurrent ovarian cancer, their caregiver, and their providers to assist in and study the decision-making process that surrounds end-of-life decisions, specifically, opting for palliative care and/or entry into hospice care. We will randomize the women and their caregivers into either our intervention or control websites. All subjects will complete a battery of demographic, psychosocial, health status and outcomes, health information, and decision making measures at baseline and 60-day post-baseline.

Once the participant has completed the baseline survey, he/she will be automatically brought to their assigned website. Both the patient and their caregiver will be assigned the same group (intervention or control). All participants will have open access to their respective study websites for a minimum of 60 days. During enrollment, participants will agree to access their respective websites at least 2-3 times per week. Both patients and caregivers assigned to the control arm will view a website containing documents generally provided as part of the usual care. They will be requested to log in with the same frequency as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Women with Stage III, IV or recurrent ovarian, primary peritoneal or fallopian tube cancer or a nominated caregiver or such women
* 18 years old or older
* At least a 5th grade education
* Able to read and write in English
* Access to computer and internet
* Voluntary written informed consent before study entry, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* No known major psychiatric or neurological diagnosis (schizophrenia or active chemical dependency)

Exclusion Criteria:

* Borderline ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Number of Women Who Completed Advanced Directive | Day 60 After Baseline
  Count of number of women with ovarian cancer who completed a new or updated their Advanced Directive during the study period.

SECONDARY OUTCOMES:
Comparison of Number of Women Who Report Appointment with Palliative Care | Day 60 After Baseline
  Count of number of women with ovarian cancer who report an appointment with a Palliative Care specialist

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A. Geller, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States